CLINICAL TRIAL: NCT01990131
Title: Suicide Risk Prevention Among Patients With Anxiety Psychopathology
Brief Title: Computerized Anxiety Treatment for Suicide
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RF02397
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Anxiety; Suicide
Keywords: computerized intervention; cognitive bias modification; anxiety; suicide
MeSH Terms: conditions — Anxiety Disorders; Suicide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The anxiety risk reduction condition will be a combination of psychoeducation plus Cognitive Bias Modification (CBM-I) for anxiety sensitivity (AS). The psychoeducational component will focus on the nature of stress and its effect on the body. Interoceptive exposure (IE) exercises, designed to correct the conditioned fear to these bodily sensations, will be explained and practiced.
  Interventions: Other: Cognitive Anxiety Sensitivity Treatment
- Control (Placebo Comparator): The control condition will be a combination of information about general health and wellness (e.g. diet, exercise etc.) plus an inert Cognitive Bias Modification (CBM-I) task.
  Interventions: Other: Physical Health Education Training

INTERVENTIONS:
Other: Cognitive Anxiety Sensitivity Treatment
  Other Names: Computerized Anxiety Treatment for Suicide (CATS)
  Arms: Intervention
Other: Physical Health Education Training
  Arms: Control

SUMMARY:
The purpose of this study is to test the effectiveness and usability of multiple computer-based treatments for mood and anxiety relevant risk factors. The target of the treatment is related to cognitive stress, which has been shown to be associated with a variety of negative mental health outcomes such as Post-Traumatic Stress Disorder, suicidal ideation, and substance use disorders.

DETAILED DESCRIPTION:
CATS is a newly developed computerized treatment targeting specific risk factors associated with anxiety symptoms and suicidal thoughts. Individuals will be asked to complete four appointments, where they will complete various self-report questionnaires as well as a newly developed computerized treatment targeting risk factors associated with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for a primary Axis 1 anxiety disorder or meet diagnostic criteria for a unipolar mood disorder along with an Axis 1 anxiety disorder.
* Show evidence of current suicidal ideation (BSS above 6.
* Show elevated AS indicated by scoring at or above the community sample mean on the ASI-Cog (above 9.

Exclusion Criteria:

* No significant medical illness (e.g. sig cardiovascular disease, epilepsy, stroke).
* Current or past psychotic-spectrum disorders or uncontrolled bipolar disorder
* No current substance dependence
* Must be an English speaker.
* Must be 18 years or older.
* Must have normal or corrected vision
* Cannot begin treatment/therapy within 1 month of baseline.
* Cannot begin a new medication within 3 months of baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 (ASI-3) | Month 4 follow-up
  The ASI-3 is an 18-item self-report measure of anxiety sensitivity (AS). This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the original ASI provides. Each subfactor is represented by six items. The measure has shown good psychometric properties.

SECONDARY OUTCOMES:
Beck Suicide Scale (BSS) | Month 4 follow-up
  The BSS is a 21-item widely used self-report measure assessing a broad spectrum of behaviors and attitudes related to suicide risk, including suicidal ideation and past suicide attempts. It has demonstrated strong reliability and validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Schmidt NB, Norr AM, Allan NP, Raines AM, Capron DW. A randomized clinical trial targeting anxiety sensitivity for patients with suicidal ideation. J Consult Clin Psychol. 2017 Jun;85(6):596-610. doi: 10.1037/ccp0000195. Epub 2017 Mar 13. PMID 28287798